CLINICAL TRIAL: NCT03847870
Title: Background Seroprevalence of Rickettsial Infections in Myanmar
Brief Title: Rickettsiae in Myanmar
Acronym: Rickettsiae
Status: Completed | Type: Observational
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: National Health Laboratory, Myanmar (Unknown); Magway General Hospital, Magway (Unknown); Monywa Hospital, Sagaing (Unknown); Mandalay General Hospital and University of Medicine, Mandalay (Unknown); University of Medicine, Magway (Unknown); Mahidol Oxford Tropical Medicine Research Unit (Other); Medical Action Myanmar (Other)
Responsible Party: Sponsor
Other Study IDs: OXTREC 552-18
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Rickettsiae Infections
Keywords: rickettsiae; seroprevalence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MORU in-house ELISA test followed by IFA if positive — An in-house rickettsial IgG ELISA test will be used for this study to determine previous rickettsial infections by measuring IgG levels. All specimens will be tested for IgG antibodies using ELISA tests for scrub typhus (Orientia tsutsugamushi strains Karp, Kato, Gilliam and TA716), murine typhus (Rickettsia typhi strain type Wilmington), and spotted fever rickettsiosis (Rickettsia honei and Rickettsia conorii). If the sample tests positive, it will be retested for the same antigens using the IFA test. The sample will be considered positive if both the ELISA and the IFA are positive.

SUMMARY:
Rickettsial infections have been found to be the second most common cause of non-malarial febrile illness in Southeast Asia, just after dengue, and are largely neglected treatable causes of morbidity and mortality. The rickettsiae can be divided into three major groups: the scrub typhus group (STG), the typhus group (TG) and the spotted fever group (SFG). Rickettsial infections typically present with an acute fever and are difficult to diagnose due to the many different causes of undifferentiated fever in Southeast Asia. Rickettsial IgG seroprevalence, reflecting past infection, will give an estimate of the burden of rickettsial infections in the population. Background seroprevalence studies in countries around Myanmar have found high rates of rickettsial infections. Yet, in Myanmar there have been no prevalence studies on rickettsial infections since the Second World War. We plan to determine IgG levels to the three different groups of rickettsial infections in leftover blood samples in several clinics and hospitals in different regions of Myanmar.

DETAILED DESCRIPTION:
Rickettsial infections have been found to be the second most common cause of non-malarial febrile illness in Southeast Asia, just after dengue, and are largely neglected treatable causes of morbidity and mortality. The rickettsiae can be divided into three major groups: the scrub typhus group (STG), the typhus group (TG) and the spotted fever group (SFG). Rickettsial infections typically present with an acute fever and are difficult to diagnose due to the many different causes of undifferentiated fever in Southeast Asia. Rickettsial IgG seroprevalence, reflecting past infection, will give an estimate of the burden of rickettsial infections in the population. The current best test for IgG serological diagnosis of previous rickettsial infections is the indirect immunofluorescence assay (IFA). IFA has several limitations

in that it is difficult to standardize due to operator subjectivity, it needs appropriate local diagnostic cut- offs and requires improvement in terms of standardization and ease of use. An alternative serological test that is cheaper and is easier to use is the enzyme-linked immunosorbent assay (ELISA), which is more suited to screen for the burden of rickettsial diseases in low-resource countries. Background seroprevalence studies in countries around Myanmar have found high rates of rickettsial infections. Yet, in Myanmar there have been no prevalence studies on rickettsial infections since the Second World War. We plan to determine IgG levels to the three different groups of rickettsial infections in leftover blood samples in several clinics and hospitals in different regions of Myanmar. Participants with leftover blood samples after having undergone a blood draw for any clinical reason or a blood donation will be requested to participate in the study. The participant will be informed about the study and requested to provide informed consent when agreeing to participate. The leftover sample will be anonymized and frozen. The gender, age and location of clinic/hospital of the participant will be recorded. All samples will be tested for IgG antibodies using an in-house ELISA test in the Mahidol Oxford Tropical Medicine Research Unit (MORU), Bangkok, Thailand for scrub typhus (Orientia tsutsugamushi strains Karp, Kato, Gilliam and TA716), murine typhus (Rickettsia typhi strain type Wilmington), and spotted fever rickettsioses (Rickettsia honei and Rickettsia conorii). If the sample tests positive for IgG antibodies, an IFA test will be performed as the gold standard reference test to confirm the finding. The anonymous samples will be discarded as soon as they are no longer needed for the study. The population investigated will be 700 patients attending seven different clinics and hospitals in different regions of Myanmar with each site including 100 patients.

We will include patients at the following study sites:

1. Himalaya general clinic, Puta-O, Kachin;
2. Lily general clinic, Thanbyuzayat, Mon;
3. Orchid general clinic, Hlaing Thar Yar, Yangon;
4. Winka general clinic, Winka, Kayin;
5. Monywa Hospital, Sagaing;
6. Mandalay General Hospital and University of Medicine, Mandalay;
7. Magway General Hospital, Magway This is a minimal risk study. The participants will not have to undergo any additional procedures, since we will be using leftover blood samples that have been collected for routine clinical tests to study the background levels of previous rickettsial infections. Participation in this study is voluntary. Subjects who decline to participate will have no impact on the care they receive at the hospital or clinic. There will be no incentives or compensation for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, all age groups, requiring a blood draw for a routine clinical purpose

Exclusion Criteria:

* Leftover blood sample of less than 500μL

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population investigated will be patients who had a leftover samples from routine clinical blood draw when attending seven different Medical Action Myanmar (MAM) clinics and hospitals in different regions of Myanmar with each site including approximately 100 patients.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Positive ELISA confirmed by positive IFA | January, 2020
  Proportion of patients with a positive IgG ELISA, subsequently confirmed with IFA, for scrub typhus (Orientia tsutsugamushi strains Karp, Kato, Gilliam and TA716), murine typhus (Rickettsia typhi strain type Wilmington), and spotted fever rickettsiosis (Rickettsia honei and Ricketsia conorii).

SECONDARY OUTCOMES:
Patient characteristics associated with rickettsial infections | January, 2020
  Correlation of different patient characteristics with a positive ELISA and IFA test indicating a previous rickettsial infection.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Anne Ashley, Dr, Principal Investigator — Myanmar Oxford Clinical Research Unit; Stuart Blacksell, Prof, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit; Philip Elders, MSc, Study Director — Myanmar Oxford Clinical Research Unit; Wei Yan Aung Htay, Dr, Study Director — Myanmar Oxford Clinical Research Unit; Yin Yin Htwe, Dr, Study Director — National Health Laboratory, Myanmar; Myat Myat Moe, Dr, Study Director — Magway General Hospital, Magway; Wai Mon Kyaw, Dr, Study Director — Monywa Hospital, Sagaing; Ni Ni Zaw, Dr, Study Director — Mandalay General Hospital and University of Medicine, Mandalay; Win May Thein, Prof, Study Director — Mandalay General Hospital and University of Medicine, Mandalay; Thin Thin Nwe, Prof, Study Director — University of Medicine, Magway; Kyaw Soe, BSc, Study Director — Myanmar Oxford Clinical Research Unit; Ampai Tanganuchitcharnchai, BSc, Study Director — Mahidol Oxford Tropical Medicine Research Unit; Ni Ni Tun, Dr, Study Director — Myanmar Oxford Clinical Research Unit and Medical Action Myanmar; Frank Smithuis, Prof, Study Director — Myanmar Oxford Clinical Research Unit and Medical Action Myanmar
Locations (1):
- Myanmar Oxford Clinical Research Unit, Yangon, Burma

REFERENCES:
- [Background] Acestor N, Cooksey R, Newton PN, Menard D, Guerin PJ, Nakagawa J, Christophel E, Gonzalez IJ, Bell D. Mapping the aetiology of non-malarial febrile illness in Southeast Asia through a systematic review--terra incognita impairing treatment policies. PLoS One. 2012;7(9):e44269. doi: 10.1371/journal.pone.0044269. Epub 2012 Sep 6. PMID 22970193
- [Background] Aung AK, Spelman DW, Murray RJ, Graves S. Rickettsial infections in Southeast Asia: implications for local populace and febrile returned travelers. Am J Trop Med Hyg. 2014 Sep;91(3):451-60. doi: 10.4269/ajtmh.14-0191. Epub 2014 Jun 23. PMID 24957537
- [Background] Trung NV, Hoi LT, Thuong NTH, Toan TK, Huong TTK, Hoa TM, Fox A, Kinh NV, van Doorn HR, Wertheim HFL, Bryant JE, Nadjm B. Seroprevalence of Scrub Typhus, Typhus, and Spotted Fever Among Rural and Urban Populations of Northern Vietnam. Am J Trop Med Hyg. 2017 May;96(5):1084-1087. doi: 10.4269/ajtmh.16-0399. PMID 28500808
- [Background] Walker DH. Rickettsial diseases in travelers. Travel Med Infect Dis. 2003 Feb;1(1):35-40. doi: 10.1016/S1477-8939(03)00025-5. PMID 17291879
- [Background] PicKard AL, McDaniel P, Miller RS, Uthaimongkol N, Buathong N, Murray CK, Telford SR 3rd, Parola P, Wongsrichanalai C. A study of'febrile illnesses on the Thai-Myanmar border: predictive factors of rickettsioses. Southeast Asian J Trop Med Public Health. 2004 Sep;35(3):657-63. PMID 15689083
- [Background] Saraswati K, Day NPJ, Mukaka M, Blacksell SD. Scrub typhus point-of-care testing: A systematic review and meta-analysis. PLoS Negl Trop Dis. 2018 Mar 26;12(3):e0006330. doi: 10.1371/journal.pntd.0006330. eCollection 2018 Mar. PMID 29579046
- [Background] Bonell A, Lubell Y, Newton PN, Crump JA, Paris DH. Estimating the burden of scrub typhus: A systematic review. PLoS Negl Trop Dis. 2017 Sep 25;11(9):e0005838. doi: 10.1371/journal.pntd.0005838. eCollection 2017 Sep. PMID 28945755
- [Background] Taylor AJ, Paris DH, Newton PN. A Systematic Review of Mortality from Untreated Scrub Typhus (Orientia tsutsugamushi). PLoS Negl Trop Dis. 2015 Aug 14;9(8):e0003971. doi: 10.1371/journal.pntd.0003971. eCollection 2015. PMID 26274584
- [Background] Civen R, Ngo V. Murine typhus: an unrecognized suburban vectorborne disease. Clin Infect Dis. 2008 Mar 15;46(6):913-8. doi: 10.1086/527443. PMID 18260783
- [Background] Uchiyama T. Tropism and pathogenicity of rickettsiae. Front Microbiol. 2012 Jun 25;3:230. doi: 10.3389/fmicb.2012.00230. eCollection 2012. PMID 22737150
- [Background] Phimda K, Hoontrakul S, Suttinont C, Chareonwat S, Losuwanaluk K, Chueasuwanchai S, Chierakul W, Suwancharoen D, Silpasakorn S, Saisongkorh W, Peacock SJ, Day NP, Suputtamongkol Y. Doxycycline versus azithromycin for treatment of leptospirosis and scrub typhus. Antimicrob Agents Chemother. 2007 Sep;51(9):3259-63. doi: 10.1128/AAC.00508-07. Epub 2007 Jul 16. PMID 17638700
- [Background] Blacksell SD, Lim C, Tanganuchitcharnchai A, Jintaworn S, Kantipong P, Richards AL, Paris DH, Limmathurotsakul D, Day NPJ. Optimal Cutoff and Accuracy of an IgM Enzyme-Linked Immunosorbent Assay for Diagnosis of Acute Scrub Typhus in Northern Thailand: an Alternative Reference Method to the IgM Immunofluorescence Assay. J Clin Microbiol. 2016 Jun;54(6):1472-1478. doi: 10.1128/JCM.02744-15. Epub 2016 Mar 23. PMID 27008880
- [Background] Phetsouvanh R, Thojaikong T, Phoumin P, Sibounheuang B, Phommasone K, Chansamouth V, Lee SJ, Newton PN, Blacksell SD. Inter- and intra-operator variability in the reading of indirect immunofluorescence assays for the serological diagnosis of scrub typhus and murine typhus. Am J Trop Med Hyg. 2013 May;88(5):932-936. doi: 10.4269/ajtmh.12-0325. Epub 2013 Mar 11. PMID 23478577
- [Background] Blacksell SD, Bryant NJ, Paris DH, Doust JA, Sakoda Y, Day NP. Scrub typhus serologic testing with the indirect immunofluorescence method as a diagnostic gold standard: a lack of consensus leads to a lot of confusion. Clin Infect Dis. 2007 Feb 1;44(3):391-401. doi: 10.1086/510585. Epub 2007 Jan 3. PMID 17205447
- [Background] Blacksell SD, Tanganuchitcharnchai A, Nawtaisong P, Kantipong P, Laongnualpanich A, Day NP, Paris DH. Diagnostic Accuracy of the InBios Scrub Typhus Detect Enzyme-Linked Immunoassay for the Detection of IgM Antibodies in Northern Thailand. Clin Vaccine Immunol. 2015 Dec 9;23(2):148-54. doi: 10.1128/CVI.00553-15. Print 2016 Feb. PMID 26656118
- [Background] Blacksell SD, Kingston HWF, Tanganuchitcharnchai A, Phanichkrivalkosil M, Hossain M, Hossain A, Ghose A, Leopold SJ, Dondorp AM, Day NPJ, Paris DH. Diagnostic Accuracy of the InBios Scrub Typhus Detect ELISA for the Detection of IgM Antibodies in Chittagong, Bangladesh. Trop Med Infect Dis. 2018 Sep 1;3(3):95. doi: 10.3390/tropicalmed3030095. PMID 30274491
- [Background] Lim C, Paris DH, Blacksell SD, Laongnualpanich A, Kantipong P, Chierakul W, Wuthiekanun V, Day NP, Cooper BS, Limmathurotsakul D. How to Determine the Accuracy of an Alternative Diagnostic Test when It Is Actually Better than the Reference Tests: A Re-Evaluation of Diagnostic Tests for Scrub Typhus Using Bayesian LCMs. PLoS One. 2015 May 29;10(5):e0114930. doi: 10.1371/journal.pone.0114930. eCollection 2015. PMID 26024375
- [Background] Pote K, Narang R, Deshmukh P. Diagnostic performance of serological tests to detect antibodies against acute scrub typhus infection in central India. Indian J Med Microbiol. 2018 Jan-Mar;36(1):108-112. doi: 10.4103/ijmm.IJMM_17_405. PMID 29735837
- [Background] Rawat V, Singh RK, Kumar A, Singh Y, Chaturvedi P, Saxena SR, Varshney U. Diagnostic validation of IgM and IgG ELISA and real-time PCR in detecting scrub typhus infection in endemic regions. J Vector Borne Dis. 2018 Apr-Jun;55(2):165-167. doi: 10.4103/0972-9062.242565. No abstract available. PMID 30280716
- [Background] Yang SL, Tsai KH, Chen HF, Luo JY, Shu PY. Evaluation of Enzyme-Linked Immunosorbent Assay Using Recombinant 56-kDa Type-Specific Antigens Derived from Multiple Orientia tsutsugamushi Strains for Detection of Scrub Typhus Infection. Am J Trop Med Hyg. 2019 Mar;100(3):532-539. doi: 10.4269/ajtmh.18-0391. PMID 30526730
- [Background] Tshokey T, Stenos J, Durrheim DN, Eastwood K, Nguyen C, Graves SR. Seroprevalence of rickettsial infections and Q fever in Bhutan. PLoS Negl Trop Dis. 2017 Nov 27;11(11):e0006107. doi: 10.1371/journal.pntd.0006107. eCollection 2017 Nov. PMID 29176880
- [Background] Khan SA, Bora T, Chattopadhyay S, Jiang J, Richards AL, Dutta P. Seroepidemiology of rickettsial infections in Northeast India. Trans R Soc Trop Med Hyg. 2016 Aug;110(8):487-94. doi: 10.1093/trstmh/trw052. Epub 2016 Sep 12. PMID 27618917
- [Background] Maude RR, Maude RJ, Ghose A, Amin MR, Islam MB, Ali M, Bari MS, Majumder MI, Tanganuchitcharnchai A, Dondorp AM, Paris DH, Bailey RL, Faiz MA, Blacksell SD, Day NPJ. Serosurveillance of Orientia tsutsugamushi and Rickettsia typhi in Bangladesh. Am J Trop Med Hyg. 2014 Sep;91(3):580-583. doi: 10.4269/ajtmh.13-0570. Epub 2014 Aug 4. PMID 25092819
- [Background] MACKIE TT. Observations on tsutsugamushi disease (scrub typhus) in Assam and Burma. Trans R Soc Trop Med Hyg. 1946 Aug;40:15-56. doi: 10.1016/0035-9203(46)90061-2. No abstract available. PMID 20998610
- [Background] Ellis RD, Fukuda MM, McDaniel P, Welch K, Nisalak A, Murray CK, Gray MR, Uthaimongkol N, Buathong N, Sriwichai S, Phasuk R, Yingyuen K, Mathavarat C, Miller RS. Causes of fever in adults on the Thai-Myanmar border. Am J Trop Med Hyg. 2006 Jan;74(1):108-13. PMID 16407353
- [Background] Watthanaworawit W, Turner P, Turner C, Tanganuchitcharnchai A, Richards AL, Bourzac KM, Blacksell SD, Nosten F. A prospective evaluation of real-time PCR assays for the detection of Orientia tsutsugamushi and Rickettsia spp. for early diagnosis of rickettsial infections during the acute phase of undifferentiated febrile illness. Am J Trop Med Hyg. 2013 Aug;89(2):308-310. doi: 10.4269/ajtmh.12-0600. Epub 2013 Jun 3. PMID 23732256
- [Background] McGready R, Ashley EA, Wuthiekanun V, Tan SO, Pimanpanarak M, Viladpai-Nguen SJ, Jesadapanpong W, Blacksell SD, Peacock SJ, Paris DH, Day NP, Singhasivanon P, White NJ, Nosten F. Arthropod borne disease: the leading cause of fever in pregnancy on the Thai-Burmese border. PLoS Negl Trop Dis. 2010 Nov 16;4(11):e888. doi: 10.1371/journal.pntd.0000888. PMID 21103369